CLINICAL TRIAL: NCT00122668
Title: Randomized Comparative Study Evaluating the Rate of Occurrence of a Lipoatrophy Syndrome in ARVnaive HIV-1 Infected Patients Receiving NRTI-Sparing Antiretroviral Regimen (Hippocampe - ANRS 121)
Brief Title: Evaluation of the Occurrence of Lipoatrophy in HIV-1 Infected Naive Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS121 HIPPOCAMPE
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections; HIV-Associated Lipodystrophy Syndrome
Keywords: HIV Protease Inhibitors; HIV-Associated Lipodystrophy Syndrome; HIV infections
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome | interventions — Protease Inhibitors

INTERVENTIONS:
Drug: non-nucleoside reverse transcriptase inhibitors
Drug: nucleoside reverse transcriptase inhibitors
Drug: protease inhibitor

SUMMARY:
The aim of this randomized study is to compare the occurrence of lipoatrophy in HIV-1 infected, naive patients receiving either a nucleoside reverse transcriptase inhibitor (NRTI)-sparing antiretroviral therapy with non-nucleoside reverse transcriptase inhibitor (NNRTI) and boosted protease inhibitor (PI), or a standard antiretroviral therapy with 2 NRTI plus either PI or NNRTI. Lipoatrophy is evaluated by measurement of fat volume by computed tomography (CT)-scan and DEXA (Dual Energy X-ray Absorptiometry).

DETAILED DESCRIPTION:
The study compare the rate of occurrence of lipoatrophy in ARVnaive HIV-1 infected patients receiving either a NRTI-sparing antiretroviral therapy with NRTI and boosted PI,or a standard antiretroviral therapy with 2 NRTI plus PI or NNRTI.

Patients were randomized (2:1:1) to either PI+NNRTI (Gp1) or standard therapy, 2NRTI+ either PI (Gp2) or + NNRTI (Gp3). The study-treatment were lopinavir/r 100/400mg bid or indinavir/r 100/400mg bid for PI-class, for NNRTI-class, efavirenz or nevirapine and all NRTIs except D4T and DDC at usual dosage.

Lipoatrophy is evaluated by evolution of subcutaneous fat in the limbs measured by DEXA (Dual Energy X-ray Absorptiometry)and CT-scan of the thighs between baseline and W96.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1-infected diagnosis
* Naive of antiretroviral treatment
* Plasma viral load (VL) over 5000 copies/ ml
* CD4 count below or equal to 350/mm3 or CD4 over 350/mm3 and VL over or equal to 100 000 copies/ml
* Written, informed consent after approval by the local human research ethics committee

Exclusion Criteria:

* Acute opportunistic infection
* Pregnancy or breast feeding
* Cytotoxic systemic chemotherapy except for Kaposi sarcoma
* Patient infected with B or C hepatitis requiring specific treatment at the beginning of the study
* Polynuclear neutrophils below 750/mm3
* Hemoglobin below 8 g/dl
* Platelets below 20 000/mm3
* Creatinine level over 1.5 (upper normal) UN
* ASAT, ALAT, bilirubin level over 3 UN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2003-11; Study Completion 2005-07

PRIMARY OUTCOMES:
Evolution of subcutaneous fat in the limbs measured by DEXA and CT-scan of the thighs between baseline and Week 96

SECONDARY OUTCOMES:
During the study until 96 weeks
Viro-immunologic efficacy: Proportion of patients with a plasma viral load below 400 and 50 copies/ml
Evolution of viral load
Evolution of CD4 lymphocytes
Evaluation of clinical safety
Evaluation of lipohypertrophic syndrome
Evaluation of glucidic and lipids metabolic profile
Evaluation of mitochondrial toxicity
Evaluation of bone toxicity by measurement of bone density
Evaluation of plasma trough concentration of protease inhibitors and non nucleoside reverse transcriptase inhibitors
Evaluation of intracellular concentration of nucleoside reverse transcriptase inhibitors
Evolution of quality of life using the World Health Organization Quality of Life in persons with HIV Brief Form (WHO-QOL-HIV BREF)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Duvivier, MD, Principal Investigator — Service des Maladies infectieuses et Tropicales, Hopital Pitie Salpetriere, Paris; Dominique Costagliola, Study Chair — INSERM U 720
Locations (1):
- Service des Maladies infectieuses et Tropicales Hopital Pitie Salpetriere, Paris, France

REFERENCES:
- [Derived] Soulie C, Assoumou L, Ghosn J, Duvivier C, Peytavin G, Ait-Arkoub Z, Molina JM, Costagliola D, Katlama C, Calvez V, Marcelin AG. Nucleoside reverse transcriptase inhibitor-sparing regimen (nonnucleoside reverse transcriptase inhibitor + protease inhibitor) was more likely associated with resistance comparing to nonnucleoside reverse transcriptase inhibitor or protease inhibitor + nucleoside reverse transcriptase inhibitor in the randomized ANRS 121 trial. AIDS. 2009 Jul 31;23(12):1605-8. doi: 10.1097/QAD.0b013e32832d9031. PMID 19487903
- [Derived] Duvivier C, Kolta S, Assoumou L, Ghosn J, Rozenberg S, Murphy RL, Katlama C, Costagliola D; ANRS 121 Hippocampe study group. Greater decrease in bone mineral density with protease inhibitor regimens compared with nonnucleoside reverse transcriptase inhibitor regimens in HIV-1 infected naive patients. AIDS. 2009 Apr 27;23(7):817-24. doi: 10.1097/QAD.0b013e328328f789. PMID 19363330
- [Derived] Duvivier C, Ghosn J, Assoumou L, Soulie C, Peytavin G, Calvez V, Genin MA, Molina JM, Bouchaud O, Katlama C, Costagliola D; ANRS 121 study group. Initial therapy with nucleoside reverse transcriptase inhibitor-containing regimens is more effective than with regimens that spare them with no difference in short-term fat distribution: Hippocampe-ANRS 121 Trial. J Antimicrob Chemother. 2008 Oct;62(4):797-808. doi: 10.1093/jac/dkn278. Epub 2008 Jul 18. PMID 18641035